CLINICAL TRIAL: NCT03477149
Title: EASYX-1 : A Multicenter Study on Safety and Efficacy of Easyx Liquid Embolization Agent Used in Five Separate Indications
Acronym: EASYX-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Antia Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K170403J; 2017-A02370-53 (Other: EUDRACT number)
Record Dates: First submitted 2018-03-09; First posted 2018-03-26 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Varicocele; Endoleak; Portal Vein Thrombosis; Bleeding; Angiomyolipoma
Keywords: liquid embolics
MeSH Terms: conditions — Varicocele; Endoleak; Hemorrhage; Angiomyolipoma

STUDY DESIGN:
Intervention Model Description: French multicenter, phase 2b (device), prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization with Easyx (Experimental): Patients requiring embolization of varicocele, portal vein before ablation, type 2 endoleak, angiomyolipoma or active bleeding will be treated with the liquid embolic agent Easyx during index procedure.
  Interventions: Device: Easyx

INTERVENTIONS:
Device: Easyx — Embolization will be done with Easyx liquid agent.

SUMMARY:
The EASYX™ Liquid Embolic is a new injectable, precipitating polymeric agent for the obliteration of vascular spaces through direct puncture or catheter access performed under X-ray guidance. The embolic liquid is an iodinized Polyvinyl Alcohol (PVA) Polymer ether. Iodine groups are covalently grafted to the PVA polymer backbone, whereby a stable nondegradable polymer with the desired features is created. The resulting polymer is dissolved in Dimethyl Sulfoxide (DMSO). EASYX™ is CE-marked since December 2016 and has been used in humans a few time for type II endoleaks, portal vein and varicocele (<10 cases at the date of submission). The purpose of this study is to evaluate the safety and efficacy of EASYX™ embolization liquid for the percutaneous treatment of vascular lesions, i.e. embolization of varicocele, type II endoleaks, portal vein before surgery, active peripheral bleeding or angiomyolipoma (AML).

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with indication of varicocele, type II endoleaks, portal vein, AML or active embolization with a liquid agent
* Aged ≥ 18 years
* Affiliated to a French health insurance system

Exclusion Criteria:

* Hypersensitivity to Polyvinyl Alcohol (PVA) Polymer
* Hypersensitivity to DMSO solvent
* Patient unable or unwilling to provide a written informed consent
* Patient participating in another interventional study
* Pregnant or breastfeeding woman
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Safety:Total number of per-procedure Serious Adverse Events (SAE) for the safety | one day
  Expected and unexpected per-procedure (SAE) related to the EASYX™ use (imputability "certain" or "probable")
Efficacy for type 2 endoleaks embolization | 6 months
  Percentage of clinical success. The clinical success of type II endoleaks embolization is defined as the stability or reduction of aneurysm's both anterioposterior and transverse diameters assessed on CT-scan at 6 months compared to baseline (4mm threshold).
Efficacy for portal vein embolization | Before ablation
  Percentage of clinical success before ablation for portal vein embolization. The clinical success of portal vein embolization is defined as the growth ≥15 % of the remnant liver assessed on presurgical CT-scan compared to baseline
Efficacy for varicocele embolization | 1 month
  Percentage of clinical success for varicocele embolization The clinical success of varicocele embolization is defined as the absence of reflux on ultrasound Doppler at one month follow-up.
Efficacy for angiomyolipoma embolization | 3 month
  Percentage of clinical success for angiomyolipoma embolization. The clinical success of angiomyolipoma embolization is defined as the reduction >10% of at least one diameter on MRI or CT-scan at 3 months follow-up compared to baseline
Efficacy for active bleeding embolization | Through embolization completion
  Percentage of clinical success for active bleeding embolization The clinical success of active bleeding embolization is defined as the complete occlusion of the target vessel assessed by angiography during the index procedure

SECONDARY OUTCOMES:
SAE | up to 6 months
  Total number of SAE
AE | up to 6 months
  Total number of AE
untargeted embolization | during procedure
  Total number of untargeted embolization
unanticipated ischemia of the target organ | up to 6 months
  Total number of unanticipated ischemia of the target organ
orchi-epididymitis | up to 6 months
  Total number of secondary post-embolization orchi-epididymitis (varicocele embolization)
neural route lesion | up to 6 months
  Total number of neural root lesion (type II endoleaks)
aneurysm rupture | up to 6 months
  Total number of aneurysm rupture (type II endoleaks)
tumor rupture | up to 6 months
  Total number of tumor rupture (angiomyolipoma)
Survival | 6 months
  Survival rates
Pain | up to 6 months
  Use of Visual Analog Scale (VAS) to evaluate the pain at device injection (between 0: no pain to 10: intolerable pain)
Pain improvement | up to 6 months
  Use of Visual Analog Scale (VAS) to evaluate the painful varicocele (between 0: no pain to 10: intolerable pain)
unanticipated use of another liquid agent | during procedure
  Total number of unanticipated use of another liquid agent for embolization
technical success | end of the procedure
  Total number of procedures with immediate technical success
Easyx volume | during procedure
  Mean volume of EASYX™ used during the index procedure
Occlusion | during procedure
  Mean degree of occlusion of the target vessel(s)
Re-intervention | up to 6 months
  Total number of re-intervention for study procedure
Interventional Radiologist (IR) satisfaction | end of the procedure
  Immediate technical satisfaction questionnaire (as perceived by the Interventional Radiologist)
Clinical efficacy | up to 6 months
  Total number of embolization clinical efficacy
Other liquid embolics | end of the procedure
  Total number of procedures with a need to complete with another liquid embolic to achieve optimal result
Quality of life | up to 6 months
  Patient's quality of life (EQ-5D)
Imaging | 6 months
  Technical success at follow-up assessed on CT-scan for type II endoleaks defined as the ability for the physician to give a diagnosis (absence or minor artifacts) on imaging

CONTACTS AND LOCATIONS:
Overall Officials: Marc SAPOVAL, MD, PhD, Principal Investigator — AP-HP - Hôpital Européen Georges Pompidou; Romaric LOFFROY, MD, PhD, Principal Investigator — CHU de Dijon - Hôpital François Mitterand; Vincent VIDAL, MD, PhD, Principal Investigator — AP-HM - La Timone
Locations (1):
- AP-HP - Hopital Europeen Georges-Pompidou Paris, France, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No